CLINICAL TRIAL: NCT03065361
Title: Assessing the Handgrip Strength, Fine Motor Skills, and Hand Sensitivity of Brazilian Children and Adolescents on Hemodialysis
Brief Title: Assessing Manual Components of Brazilian Children and Adolescents on Hemodialysis
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Thais Thaler Souza, MSc, Federal University of Minas Gerais
Other Study IDs: 1.305.695
Record Dates: First submitted 2017-01-21; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Handgrip Strength; Fine Motor Skills; Sensitivity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Group composed of 21 children and adolescents aged between 9 and 19 years old, treated by hemodialysis in two hospitals of Belo Horizonte. Just in case of some evidence of difference in the results within group A, because of the two types of dialysis (via fistula or catheter), this group can be subdivided in subgroups A1 (n=10) and A2 (n=11), respectively.
  Group A was already on hemodialysis, the intervention was not performed by the researcher. Our goal was only to evaluate some characteristics of these individuals.
- Group B: Group composed of 21 children and adolescents matching age and gender for the Group A participants. The individuals were recruited in schools of Belo Horizonte.

SUMMARY:
The purpose of this study was to assess the handgrip strength; fine motor skills; and hand sensitivity of Brazilian children and adolescents with Chronic Kidney Diseases (CKD). The sample was composed by 42 children and adolescents, 21 on hemodialysis (group A) and the other 21 acted as the control group (group B). The performance of both groups was compared. The outcome measures included Jebsen-Taylor Hand Function Test, the Semmes Weinstein monofilaments test and Jamar Dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CKD with active hemodialysis treatment (only to group A);
* Ability to understand the tests and questionnaires applied.

Exclusion Criteria:

* Neuropsychiatric disease associated; and
* Any medical contraindication against the participation in the study.

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The participants of the group A were not randomized children and adolescents performing hemodialysis treatment in two hospitals of Belo Horizonte. Findings obtained in patients were compared to children and adolescents matched by age and sex, which participants were recruited in schools of Belo Horizonte and metropolitan region part of the group B.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Jebsen-Taylor Hand Function Test | 30 minutes
  The manual functioning of upper limbs were assessed by the Jebsen-Taylor Hand Function Test, a standardized test composed by manual tasks based on daily activities. The test is divided into seven sub-tests: (1) writing, (2) flipping cards, (3) small objects lifting, (4) spoon usage, (5) blocks stacking, (6) large and lightweight objects lifting, and (7) large and heavy objects lifting.

SECONDARY OUTCOMES:
The Semmes Weinstein Monofilaments Test | 10 minutes
  The Semmes Weinstein monofilaments test was used to evaluate the skin threshold sensitivity. In this test, the damage to the skin sensitivity is classified in colors. The eyes are blindfolded and the nylon monofilaments are applied to the hands of participants until the touch is felt in the dermatomes, regarding the distribution of the ulnar, median and radial.
Jamar Dynamometer | 15 minutes
  The handgrip strength was checked by the Jamar® Dynamometer, it is constituted by a voltage sealers system which indicates on the device the handgrip strength in kilograms/strength (kg/f) or in pounds/inch. The device was used three times before and after hemodialysis session, and the results were based on the average of the three applications. In the group B, the test was applied 3 times, and obtained average. The dynamometer works in many situations in order to determine the functionality of the hands and is considered a "gold standard" for this purpose.

OTHER OUTCOMES:
Edinburgh Handedness Inventory | 15 minutes
  The handedness setting was defined by the Edinburgh Handedness Inventory,

CONTACTS AND LOCATIONS:
Overall Officials: Thais T Souza, MSc, Principal Investigator — Federal University of Minas Gerais

IPD SHARING:
Plan to Share IPD: Undecided